CLINICAL TRIAL: NCT06441578
Title: Special Drug Use Surveillance of ADZYNMA Intravenous 1500 (All-Case Investigation)
Brief Title: A Survey of Recombinant ADAMTS13 in Participants With Congenital Thrombotic Thrombocytopenic Purpura
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-755-4005; jRCT2031240130 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recombinant ADAMTS13: Participants will receive recombinant ADAMTS13 intravenous injection.
  Interventions: Drug: Recombinant ADAMTS13

INTERVENTIONS:
Drug: Recombinant ADAMTS13 — Recombinant ADAMTS13, Intravenous injection
  Other Names: ADZYNMA Intravenous 1500; TAK-755

SUMMARY:
This study is a survey in Japan of recombinant ADAMTS13 used to treat or to prevent participants with congenital thrombotic thrombocytopenic purpura (cTTP). The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects related from recombinant ADAMTS13 and to check if recombinant ADAMTS13 improves or prevents cTTP.

During the study, participants with cTTP will take recombinant ADAMTS13 intravenous injection according to their clinic's standard practice. The study doctors will check for side effects from recombinant ADAMTS13 for 18 months.

ELIGIBILITY:
Inclusion Criteria:

- All participants with congenital thrombotic thrombocytopenic purpura (cTTP), treated with recombinant ADAMTS13

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2032-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience at Least One Treatment-Emergent Adverse Events (TEAE) | Up to 18 Months

SECONDARY OUTCOMES:
Percent Change in Observed Platelet Count from Baseline at the End of Treatment | Up to 18 Months
  Percent change in platelet count from baseline at the end of treatment will be reported.
Percent Change in Observed ADAMTS13 Activity from Baseline at the End of Treatment | Up to 18 Months
  Percent change in ADAMTS13 activity from baseline at the end of treatment will be reported.
Percent Change in Observed ADAMTS13 Inhibitor from Baseline at the End of Treatment | Up to 18 Months
  Percent change in ADAMTS13 inhibitor from baseline at the end of treatment will be reported.
Number of Participants with Thrombotic Thrombocytopenic Purpura (TTP) Events on Periodic Replacement Therapy | Up to 18 Months
  Number of participants with TTP events on periodic replacement therapy will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/c2fc7ca33be64ac7